CLINICAL TRIAL: NCT05774379
Title: The Effect of Virtual Reality and Fatigue Education on Fatigue and Anxiety Levels in Children With Cancer
Brief Title: Virtual Reality and Fatigue Education
Acronym: VRfatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gülçin Özalp Gerçeker, pHD, Assoc. Prof., Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5776GOA
Record Dates: First submitted 2023-03-07; First posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Fatigue; Anxiety
Keywords: virtual reality
MeSH Terms: conditions — Fatigue; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality and fatigue education (Experimental): watching the application by wearing virtual glasses for 3 days and Providing training on fatigue to all children (1 session, average 45 minutes) (using role-play, exercise, games, coloring books and activity materials)
  Interventions: Device: virtual reality and fatigue education
- fatigue education (Experimental): Providing training on fatigue to all children (1 session, average 45 minutes) (using role-play, exercise, games, coloring books and activity materials)
  Interventions: Behavioral: fatigue education

INTERVENTIONS:
Device: virtual reality and fatigue education — virtual reality distraction for 3 days and fatigue education for children
  Arms: virtual reality and fatigue education
Behavioral: fatigue education — fatigue education for children
  Arms: fatigue education

SUMMARY:
It was planned to evaluate the effect of distraction intervention with virtual reality and fatigue education on the level of fatigue and anxiety in children with cancer.

DETAILED DESCRIPTION:
H1: The fatigue scores of the patients who received distraction intervention with virtual reality and were given fatigue training were lower than the group that was given only fatigue training.

H2: The anxiety scores of the patients who received distraction intervention with virtual reality and were given fatigue training were lower than the group that was given only fatigue training.

Data collection After the child and his family are informed about the study, their written informed consent will be obtained. All children included in the study on the day (day 0) prior to the start of chemotherapy treatment will be given training on fatigue. In order to determine how he felt and his level of fatigue on the day of the training, it was planned to apply the Child Anxiety Scale-State (CAS-D), Child Fatigue Scale-24 Hours and Visual Fatigue Scale at 16.00 (pretest).

After randomization is achieved, a distraction intervention will be applied once a day for 10-15 minutes with virtual glasses on the 1st, 2nd and 3rd days of the chemotherapy treatment of the children in the study group. This intervention is planned to take place between 14.00-15.00 in the afternoon.

ELIGIBILITY:
Inclusion Criteria:

* Be between 7-18 years old
* Inpatient chemotherapy treatment for more than three days
* 4 weeks over the time of diagnosis (not in the induction phase)
* Having a hemoglobin level above the criteria for transfusion of blood products (8 mg/dl for hematological malignancies, below 7 mg/dl for oncological malignancies).
* The child voluntarily agrees to participate in the study and consent is obtained from the child and parent

Exclusion Criteria:

* Being in terminal period
* undergoing a surgical operation
* Unwillingness to participate in the study

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
fatigue | pretest, 1., 2. and 3. days of chemotheraphy
  Child Fatigue Scale-24 Hours: It consists of 10 items related to the perception of fatigue in children with cancer. The items in the scale contain statements that will show the child's experience of fatigue-related symptoms in the last 24 hours. The items were arranged according to likert scoring between 'never (1)' and 'a lot (5)'.
anxiety | pretest, 1., 2. and 3. days of chemotheraphy
  The Children's Anxiety Meter (CAM-S). The Children's Anxiety Meter assesses children's anxiety and uses before medical procedures. This scale is drawn like a thermometer with a bulb at the bottom and also includes horizontal lines at intervals going up to the top (0-10). This scale ranges from 0 to 10. Higher values represent higher anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Gülçin Özalp Gerçeker, pHD, RN, Principal Investigator — Dokuz Eylul University
Locations (1):
- Gülçin Özalp Gerçeker, Izmir, Turkey (Türkiye)